CLINICAL TRIAL: NCT00286585
Title: Multi-Center Trial on the Effect of Anesthetics on Morbidity and Mortality in Patients Undergoing Major Non-cardiac Surgery
Brief Title: TEAM-Project: Trial on the Effect of Anesthetics on Morbidity and Mortality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 261/05; IIS-SWIT-05-002
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: preconditioning; cardiac protection; morbidity; mortality; major non-cardiac surgery; cardiac mortality and morbidity; high cardiac perioperative risk
MeSH Terms: conditions — Coronary Artery Disease | interventions — Sevoflurane; Anesthetics, Intravenous; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhalational anesthetic (Active Comparator): Sevoflurane will be used as the main anesthetic in this arm, and no propofol will be administered
  Interventions: Drug: Inhalational anesthetic
- Intravenous anesthetic, propofol (Active Comparator): Propofol will be used as the main anesthetic in this arm, and no inhalational anesthetic will be administered
  Interventions: Drug: Intravenous anesthetic, propofol

INTERVENTIONS:
Drug: Inhalational anesthetic — Sevoflurane, dosage according to the physician in charge
  Other Names: Ultane,; Sevorane
  Arms: Inhalational anesthetic
Drug: Intravenous anesthetic, propofol — Propofol, dosage according to the physician in charge
  Other Names: Diprivan,; Diprovan
  Arms: Intravenous anesthetic, propofol

SUMMARY:
Volatile anesthetics may provide some protection from myocardial ischemia, an effect called anesthetic preconditioning. In patients undergoing coronary artery bypass surgery, this preconditioning effect resulted in better cardiac performance, faster recovery and lower morbidity and mortality.

The investigators will perform a prospective randomized multi-center study to compare volatile with total intravenous anesthesia in patients at a high cardiac risk who undergo major non-cardiac surgery.

DETAILED DESCRIPTION:
Basic research and animal studies have detected that volatile anesthetics provide some protection from myocardial ischemia, an effect called anesthetic preconditioning. Recent clinical studies have found that this preconditioning effect is of clinical relevance in patients undergoing coronary artery bypass surgery, resulting in better cardiac function and faster recovery after surgery, and in lower one-year morbidity. In patients undergoing non cardiac surgery, cardiac complications also are the major cause of perioperative morbidity and mortality. Myocardial ischemia frequently occurs during and immediately after non cardiac surgery in patients with coronary artery disease, and is a strong predictor of subsequent cardiac complications and death. Whether or not volatile anesthetics also provide clinically relevant protection from perioperative ischemia and subsequent cardiac complications in patients undergoing non cardiac surgery is unknown. Therefore, we will perform a prospective, randomized multi-center study to compare volatile with total intravenous anesthesia in patients at high cardiac risk who undergo major non cardiac surgery. We hypothesize that the use of a volatile anesthetic will reduce the incidence of perioperative ischaemia and myocardial injury, as indicated primarily by less ST-segment changes in the Holter ECG and, if there will be an effect, secondarily by lower incidences of elevated troponin T and NT-pro-BNP levels. And we hypothesize that the use of a volatile anesthetic will reduce the one-year incidence of cardiac complications and all cause mortality after surgery. The results of this study may apply to a huge percentage of surgical patients because coronary artery disease is the clinically most relevant co-morbidity, and its prevalence is expected to increase with the steadily increasing number of surgical patients aged 65 yr and older.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a non-cardiac surgical procedure of high or intermediate cardiac risk are eligible if they have documented coronary artery disease (CAD) or are at high risk of CAD.

Exclusion Criteria:

* Ongoing medication with sulfonylurea derivatives (unless stopped ≥ 2 days before surgery) or theophylline
* Emergency surgery
* Unstable angina pectoris
* Preoperative hemodynamic instability
* Severe hepatic disease
* Renal insufficiency (creatinine clearance < 30 ml/min)
* Severe chronic obstructive pulmonary disease (forced expiratory volume in 1 second [FEV1] < 1 litre)
* Absence of written patient consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2006-02; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Ischemia (Holter-electrocardiogram [ECG], troponin T, ECG) | 7 days postoperatively

SECONDARY OUTCOMES:
Congestive heart failure (N-terminal B-type natriuretic peptide [NT-pro-BNP]) | 2 days postoperatively
influence of genetic polymorphism on cardiac morbidity and mortality | 7 days, 6 and 12 months
cardiac morbidity and mortality | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Seeberger, Prof. Dr., Principal Investigator — Department of Anesthesia, University Hospital, Basel, Switzerland
Locations (3):
- Switzerland (3):
  - Kantonsspital, Liestal, Basel-Landschaft
  - University Hospital, Basel, Basel
  - Bürgerspital, Solothurn, Canton of Solothurn

REFERENCES:
- [Derived] Mauermann E, Bolliger D, Seeberger E, Puelacher C, Corbiere S, Filipovic M, Seeberger M, Mueller C, Lurati Buse G. Incremental Value of Preoperative Copeptin for Predicting Myocardial Injury. Anesth Analg. 2016 Dec;123(6):1363-1371. doi: 10.1213/ANE.0000000000001635. PMID 27870734
- [Derived] Lurati Buse GA, Schumacher P, Seeberger E, Studer W, Schuman RM, Fassl J, Kasper J, Filipovic M, Bolliger D, Seeberger MD. Randomized comparison of sevoflurane versus propofol to reduce perioperative myocardial ischemia in patients undergoing noncardiac surgery. Circulation. 2012 Dec 4;126(23):2696-704. doi: 10.1161/CIRCULATIONAHA.112.126144. Epub 2012 Nov 7. PMID 23136158